CLINICAL TRIAL: NCT01189357
Title: Revision Meniscal Transplants; Lateral and Medial
Status: Completed | Type: Observational
Sponsor: University Hospital, Ghent (Other)
Responsible Party: René Verdonk, University Hospital, Ghent
Other Study IDs: 2010/358
Record Dates: First submitted 2010-08-25; First posted 2010-08-26 (Estimated); Last update posted 2011-07-14 (Estimated); Status verified 2011-07

CONDITIONS: Revision of Meniscal Transplant
Keywords: meniscal transplant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- failed meniscal transplantation

SUMMARY:
During the period 1989-1999, a number of patients underwent a meniscal transplantation. A few transplants were not successful. These patients form the population of this study. They all underwent a Total Knee Prosthesis (TKP) or unicompartmental knee prosthesis (UKP) after the failure of the transplants The goal of this study is to evaluate their current medical condition, to perform a survival analysis, and to determine the clinical outcome.

The clinical result will be stipulated by means of standardized questionnaires (KOOS, HSS and SF-36)and clinical examination.

ELIGIBILITY:
Inclusion Criteria:

* failed Meniscal transplantation between 1989 and 1999

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: failed meniscal transplantation
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2010-10; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Perform a survival analysis of meniscal transplants. Failure of transplant was defined as replacement of the allograft by a knee prothesis. | 20 years after surgery
  The clinical result will be stipulated by means of standardized questionnaires (KOOS, HSS and SF-36) and clinical examination.

SECONDARY OUTCOMES:
Clinical evaluation of the knee after TKP/UKP following a failed meniscal transplant. | 20 years after surgery

CONTACTS AND LOCATIONS:
Overall Officials: René Verdonk, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- See also: website University Hospital Ghent — http://www.uzgent.be